CLINICAL TRIAL: NCT07105137
Title: Artificial Intelligence-Assisted Expressive Writing Intervention to Improve Adolescent Emotional Distress: A Cluster Randomized Controlled Trial
Brief Title: AI-assisted GNW on Adolescent Emotional Distress
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Yinyin Zang, PhD, Principal Investigator, Peking University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AI-assisted GNW
Record Dates: First submitted 2025-05-16; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Emotional Disturbance; Emotional Regulation; Insomnia
Keywords: AI-assisted; Expressive writing; Adolesents; Emotional distress; Insomnia
MeSH Terms: conditions — Affective Symptoms; Emotional Regulation; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: To maintain rigorous protection against bias, allocation to the AI-GNW, NF-GNW, or NWG arms was concealed from participants, interventionists, and those responsible for outcome evaluation. Participants were informed only that they would engage in a writing exercise and were unaware of the nature or content of the feedback provided in the AI-GNW arm. Investigators who facilitated the sessions did not have access to the randomization schedule or to any identifying information about group assignment. Outcomes assessors remained blind to each participant's study arm. This triple-masking procedure ensured that neither expectations nor assessment procedures could differentially influence intervention delivery or measurement of study endpoints.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AI-GNW (Experimental)
  Interventions: Behavioral: AI-GNW
- NF-GNW (Active Comparator)
  Interventions: Behavioral: NF-GNW
- NWG (Sham Comparator)
  Interventions: Behavioral: NWG

INTERVENTIONS:
Behavioral: AI-GNW — This is a three-day writing intervention. Each session lasts 20 minutes. On the first day, participants in both GNW conditions will recount a negative experience and reflect on their thoughts and feelings; on the second day, they will focus exclusively on the negative aspects of that experience; and on the third day, they will explore its positive dimensions. AI-GNW participants would receive AI-generated feedback.
  Arms: AI-GNW
Behavioral: NF-GNW — guided narrative writing without feedbacks
  Arms: NF-GNW
Behavioral: NWG — In contrast, NWG participants will objectively document their previous day's daily routine.
  Arms: NWG

SUMMARY:
This cluster-randomized controlled trial aims to evaluate the efficacy of an AI-assisted Guided Narrative Writing (AI-GNW) in alleviating emotional distress among adolescents. Classes will be randomized in a 1:1:1 ratio to one of three arms-AI-GNW, a no-feedback GNW (NF-GNW), or a Neutral Writing Group (NWG)-and will complete a three-day writing intervention. On the first day, participants in both GNW conditions will recount a negative experience and reflect on their thoughts and feelings; on the second day, they will focus exclusively on the negative aspects of that experience; and on the third day, they will explore its positive dimensions. In contrast, NWG participants will objectively document their previous day's daily routine. After each session, those in the AI-GNW arm will receive individualized, AI-generated feedback, whereas NF-GNW participants will proceed without feedback.

DETAILED DESCRIPTION:
Adolescent mental health, and in particular emotional distress, has emerged as a global public health challenge. A recent meta-analysis of 80,879 adolescents found that approximately 25.2 percent experienced clinically significant depression and 20.5 percent suffered from anxiety, with these emotional disturbances accounting for an estimated 45 percent of the total disease burden in this age group. In China, the situation is equally alarming: the 2022 Blue Book on National Depression reports that roughly half of all individuals diagnosed with an emotional disorder are school-aged, and as many as 41 percent have interrupted their studies as a result. Beyond inflicting serious harm on adolescents' physical and psychological well-being, persistent emotional distress undermines social engagement and academic performance, and may precipitate more severe psychopathology, such as major depression, anxiety disorders, or even suicidal behaviors, placing a heavy burden on families, communities, and the public health system. Thus, early and effective intervention is of paramount importance for improving youth mental health.

Schools represent a central arena in adolescents' daily lives and an ideal platform for delivering psychological interventions. In response to rising rates of youth emotional problems, the Chinese government has enacted a series of policies to bolster mental health education and intervention in schools. However, the vast size of China's adolescent population and the relative scarcity of professional resources mean that traditional one-to-one intervention models have limited reach when implemented at scale. Many schools lack sufficient numbers of qualified counselors, and non-specialist teachers often do not possess the training needed to deliver sustained, targeted support, resulting in modest and non-durable effects on students' emotional well-being.

Moreover, school-based intervention programs confront several practical challenges. First, the number of licensed school-psychology professionals remains inadequate in many regions, leaving schools unable to provide consistent, high-quality support. Second, a persistent mismatch between intervention demand and available resources makes it difficult to tailor services to individual students' needs, undermining the overall effectiveness of existing programs.

Among the array of psychological interventions, writing-based approaches have gained prominence for their simplicity, low cost, and ease of dissemination in group settings such as classrooms. Writing interventions typically guide participants to articulate their emotions and thoughts in writing for 20-30 minutes per day over 3-5 consecutive days, thereby fostering emotional processing, adaptive expression, and the construction of personal meaning. Meta-analytic evidence confirms that such interventions yield significant improvements in emotional symptoms and related psychophysiological outcomes, including sleep quality. In Chinese adolescent populations, guided narrative writing has been shown to reduce examination anxiety and to ameliorate symptoms of depression and anxiety. Nevertheless, conventional writing interventions often lack mechanisms for timely, individualized feedback, which can dampen participant engagement and undermine the longevity of treatment gains.

Against this backdrop, the integration of artificial intelligence (AI) offers promising new avenues for enhancing psychological interventions. Prior research indicates that interventions incorporating ongoing, process-oriented feedback and interactive dialogue outperform those that provide no feedback. Yet, in large-scale implementations, human-delivered feedback is constrained by finite personnel resources. By leveraging natural-language processing techniques, AI systems can automatically detect emotional and cognitive markers in written text and deliver personalized feedback at scale, thereby addressing a critical gap in current practice. Introducing AI-driven feedback into adolescent writing interventions thus holds considerable promise for improving outcomes in emotional distress.

Building on these insights, the present study will recruit approximately 1,000 adolescent students and-using classes as clusters-randomly assign them in equal proportions to one of three arms: an AI-feedback Guided Narrative Writing group (AI-GNW), a no-feedback Guided Narrative Writing group (NF-GNW), or a Neutral Writing Group (NWG). We will evaluate the impact of AI-assisted narrative writing on emotional distress, comparing the trajectories of change across these three conditions.

ELIGIBILITY:
Inclusion Criteria:

* Native speakers of Chinese who are proficient in reading and writing Chinese.
* Signed a informed consent form and voluntarily agreed to participate.
* Owns a smartphone, tablet, or similar electronic device and is able to complete the required questionnaires and writing tasks.

Exclusion Criteria:

* Prior clinical diagnosis of schizophrenia or any other major psychiatric disorder.
* Presence of severe cognitive impairment, language-expression difficulties, or any other condition that would impede writing ability.
* Participation in another similar psychological intervention or psychotherapy within the past three months.
* Inability to tolerate a group-based intervention setting due to personal health conditions (e.g., serious illness).
* Unwillingness or inability to provide necessary cooperation or to sign the informed consent form.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 900 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Revised Child Anxiety and Depression Scale (RCADS) | Baseline (day 0), post-intervention (day 4), and follow-ups at 1 (day 34),3 (day 64), and 6 (day 94) months after the intervention.
  RCADS is a 25-item scale that includes 15 items for general anxiety and 10 for depression, rated on a 4-point Likert scale (0 = never, 3 = always). Higher scores mean more severe emotional distress
Insomnia Severity Index (ISI) | Baseline (day 0), post-intervention (day 4), and follow-ups at 1 (day 34),3 (day 64), and 6 (day 94) months after the intervention.
  ISI is a 7-item, 5-point (0-4) Likert scale. Higher scores mean higher insomnia severity.

SECONDARY OUTCOMES:
Non-Suicidal Self-Injury Assessment Tool (NSSI-AT) | Baseline (day 0), post-intervention (day 4), and follow-ups at 1 (day 34),3 (day 64), and 6 (day 94) months after the intervention.
  Only the severity dimension was measured in this trial.
Suicidal Behaviors Questionnaire-Revised (SBQ-R) | Baseline (day 0), post-intervention (day 4), and follow-ups at 1 (day 34),3 (day 64), and 6 (day 94) months after the intervention.
Chinese PTSD Symptom Scale (CPSS) | Baseline (day 0), post-intervention (day 4), and follow-ups at 1 (day 34),3 (day 64), and 6 (day 94) months after the intervention.

OTHER OUTCOMES:
Adverse Childhood Experience Questionnaire (ACE) | Baseline (day 0)
Beijing Irritability Scale (BIS) | Baseline (day 0), post-intervention (day 4), and follow-ups at 1 (day 34),3 (day 64), and 6 (day 94) months after the intervention.
Positive Childhood Experience Questionnaire (PCE) | Baseline (day 0)
Connor-Davidson Resilience Scale (CD-RISC) | Baseline (day 0), post-intervention (day 4), and follow-ups at 1 (day 34),3 (day 64), and 6 (day 94) months after the intervention.
Cognitive Emotion Regulation Questionnaire (CERQ) | Baseline (day 0), post-intervention (day 4), and follow-ups at 1 (day 34),3 (day 64), and 6 (day 94) months after the intervention.
  Only the Catastrophication dimension was measured in the trial.
Emotion Awareness Questionnaire (EAQ) | Baseline (day 0), post-intervention (day 4), and follow-ups at 1 (day 34),3 (day 64), and 6 (day 94) months after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University, Haidian, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
To protect participants' privacy, authors wishing to access the data should contact the corresponding author and provide a statistical analysis plan addressing a new research question. The study trial management group will discuss all requests.